CLINICAL TRIAL: NCT00615329
Title: The Huntsman Cancer Institute - The Use of Microarray Analysis in Characterizing Mesenchymal Tissue Tumors: Differentiation of Normal, Benign, and Malignant Conditions
Brief Title: Huntsman Biopsy Study
Status: Terminated | Type: Observational
Why Stopped: Huntmans Cancer Institute terminated study
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Huntsman Cancer Institute (Other)
Responsible Party: Principal Investigator, Timothy Damron, M.D., Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: Huntsman Cancer Institute; IRB 4795 (Other: IRB number)
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Soft Tissue Sarcoma; Osteosarcoma
Keywords: Create tumor specific gene profiles to improve diagnostic accuracy; Perform gene set validation for diagnostic predictive power; Define deviant gene list implicated in pathogenesis
MeSH Terms: conditions — Sarcoma; Osteosarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cDNA microarrays facilitate the systematic and comprehensive analysis of transcriptional alterations occurring in diseased tissues.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Soft tissue tumor: Any patient with soft tissue tumor will be asked to give a sample for this study

SUMMARY:
Bone and soft tissue sarcomas are currently classified based upon light microscopy supplemented by immunohistochemistry, but within many if not all of these tumor histologic types, considerable heterogeneity exists not only in microscopic appearance but also in biologic behavior and prognosis. Progress in the directed treatment of these tumors, particularly the sarcomas, awaits characterization of the gene profiles for these tumors. Orthopedic oncology researchers at Huntsman Cancer Institute at the University of Utah are establishing a tumor bank for this purpose. The long term objectives of this work include:

1. creating tumor specific gene profiles to improve diagnostic accuracy
2. performing gene set validation for diagnostic predictive power
3. defining a discriminate gene list implicated in pathogenesis

The tissue procured under this protocol at SUNY Upstate Medical University will be limited to excess soft tissue and bone tumor tissue from patients otherwise undergoing clinically indicated procedures for diagnosis or treatment under the care of the local principal investigator (PI) and will be forwarded to the central investigator, R. Lor Randall, MD at Huntsman Cancer Institute for use in the characterization of the gene profiles of these tumors.

DETAILED DESCRIPTION:
as stated in brief summary

ELIGIBILITY:
Inclusion Criteria:

* Bone or soft tissue tumor that has been established to be or is suspected to possibly be a sarcoma AND who will require a diagnostic or therapeutic surgical procedure which will result in procurement of tissue for histologic review

Exclusion Criteria:

* Non cancer patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who present to Doctor Damron for care relating to a bone or soft tissue tumor that has been established to be or is suspected to possibly be a sarcoma AND who will require a diagnostic or therapeutic surgical procedure which will result in procurement of tissue for histologic review will be approached in the consent process.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2003-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Classification of sarcomas | Upon collection/analysis of sarcoma
  sarcomas will be classified by researchers at Huntsman Institute

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Damron, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States